CLINICAL TRIAL: NCT03036826
Title: Computer-basierte Dosierungsregime Von Antiinfektiva Bei eingeschränkter Nierenfunktion Und Kontinuierlichen Nierenersatztherapieverfahren (Computer-based Dosage Calculation for Antibiotics in Patients With Impaired Renal Function or Renal Replacement Therapy)
Brief Title: Computer-based Dosage Calculation for Antibiotics
Status: Withdrawn | Type: Observational
Why Stopped: due to organisational changes
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: CADDy
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2018-10

CONDITIONS: Acute Kidney Insufficiency; Anti-Infective Agent Toxicity
Keywords: renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Piperacillin, Tazobactam Drug Combination; Meropenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Piperacillin/Tazobactam: Group of patients receiving Piperacillin/Tazobactam as antiinfective therapy
  Interventions: Drug: Piperacillin/tazobactam
- Meropenem: Group of patients receiving Meropenem as antiinfective therapy
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Piperacillin/tazobactam — antiinfective therapy with Piperacillin/Tazobactam within routine care
  Groups: Piperacillin/Tazobactam
Drug: Meropenem — antiinfective therapy with Meropenem within routine care
  Groups: Meropenem

SUMMARY:
Adequate dosing of antiinfective therapy in critically ill patients with impaired or lost renal function or continuous renal replacement therapy is nearly impossible without measuring the drug concentration in blood samples. In many hospitals that is still not an option. The investigators aim to show, that computer based calculation can avoid over- or under-dosing.

DETAILED DESCRIPTION:
Adequate dosing of antiinfective therapy in critically ill patients is most important to improve outcome. Patients with impaired or lost renal function or continuous renal replacement therapy are hard to calculate using drug information sheets or "lists" with recommendations. It is nearly impossible to avoid drug levels that are much to low or much to high without measuring the concentration in blood samples. Since that possibility is still not available in every clinic we aim to show, how a computer based calculation can help to find the adequate dosing.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring antiinfective therapy
* patients with impaired renal function or requiring continuous renal replacement therapy

Exclusion Criteria:

* plasmapheresis or liver replacement therapy
* renal replacement therapy with integrated CytoSorb®-Membrane
* extracorporal live support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients with impaired renal function and antiinfective therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
drug levels (blood) | 3 days
  achieved drug levels in blood samples

SECONDARY OUTCOMES:
dosing changes | 3 days
  dose adjustments to the computer based calculated regiments

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Prohaska, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided